CLINICAL TRIAL: NCT04216615
Title: Effect of Preoperative Anxiety on Postoperative Delirium in Elderly Patients Undergoing Orthopaedic Surgery.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Jin Dong Liu, Principal Investigator, Xuzhou Medical University
Other Study IDs: XYFY-2019-0156
Record Dates: First submitted 2019-12-31; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Delirium; Anxiety
MeSH Terms: conditions — Delirium; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with preoperative anxiety
  Interventions: Behavioral: preoperative anxiety
- patients without preoperative anxiety
  Interventions: Behavioral: preoperative anxiety

INTERVENTIONS:
Behavioral: preoperative anxiety — patients who are anxious

SUMMARY:
Postoperative delirium is a common and important complication in patients. The aim of this study was to investigate whether preoperative anxiety predicted onset of postoperative delirium in elderly patients undergoing orthopaedic surgery, so as to help develop preventive approaches.

ELIGIBILITY:
Inclusion Criteria:

* aged 65 or older
* patients undergoing elective orthopaedic surgery
* ASA I-III

Exclusion Criteria:

* history of craniocerebral trauma surgery or severe central nervous system disease
* inability to read or understand the informed consent documents
* too physically or psychologically ill

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: 290 elderly patients undergoing elective orthopaedic surgery in the Affiliated Hospital of Xuzhou Medical University.
Sampling Method: Probability Sample
Enrollment: 290 (Estimated)
Dates: Start 2020-01-04 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | 5-day postoperative period
  postoperative delirium is diagnosed using CAM

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data(IPD) will be available when this trial is finished and the article have been published.